CLINICAL TRIAL: NCT05219435
Title: Phase II Non Randomized Clinical Trial of NIVOLUMAB/IPILIMUMAB Maintenance Following First-line Chemotherapy in Unresectable Locally Advanced or Metastatic Urothelial Cancer.
Brief Title: Study of NIVOLUMAB/IPILIMUMAB Maintenance in Unresectable Locally Advanced or Metastatic Urothelial Cancer
Acronym: VEXILLUM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Oncology Genito-Urinary Group (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOGUG-2021-IEC(VEJ)-4; 2021-005364-22 (EudraCT Number)
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Urothelial Cancer
Keywords: metastatic; unresectable locally advanced
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: Patients will receive maintenance therapy with 4 cycles of Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg every three weeks (Q3W)(induction phase) followed by Nivolumab 480 mg every 4 weeks (Q4W)(consolidation phase) until unacceptable toxicity, disease progression (PD), investigator ́s decision, patient's consent withdrawal or death by any cause, whichever occurs first.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nivolumab plus Ipilimumab (Experimental): Patients will receive maintenance therapy with 4 cycles of Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg every three weeks (Q3W)(induction phase) followed by Nivolumab 480 mg every 4 weeks (Q4W)(consolidation phase) until unacceptable toxicity, disease progression (PD), investigator ́s decision, patient's consent withdrawal or death by any cause, whichever occurs first.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab at 1 mg/kg by intravenous (IV) infusion on D1 of each cycle. Nivolumab at a fixed dose of 480 mg by intravenous (IV) infusion on D1 of each cycle. The maximum duration of treatment with nivolumab will be 2 years, and patients will discontinue treatment at any time in case of unacceptable toxicity, disease progression (PD), investigator ́s decision, patient's consent withdrawal or death by any cause, whichever occurs first.
  Other Names: Opdivo
Drug: Ipilimumab — Ipilimumab at 3 mg/kg by intravenous (IV) infusion on D1 of each cycle.
  Other Names: Yervoy

SUMMARY:
Immunotherapy has improved clinical outcomes in metastatic urothelial carcinoma (mUC). Second-line treatment after progression to platinum-containing chemotherapy with immune checkpoint inhibitors (ICIs) have antitumor activity in advanced / metastatic UC and provide favorable safety profiles when compared with chemotherapy The study aims to determine if Nivolumab plus Ipilimumab maintenance therapy is effective in delaying disease progression in patients with unresectable locally advanced or metastatic urothelial cancer that did not progress during or following completion of first-line chemotherapy. Vexillum plans to recruit patients that achieve clinical benefit from first-line chemotherapy and may be candidates for maintenance immunotherapy to consolidate this benefit.

DETAILED DESCRIPTION:
All enrolled patients should have received first-line chemotherapy and not progressed. After a treatment-free interval of 3-12 weeks from chemotherapy, patients will receive maintenance therapy with 4 cycles of Nivolumab 1 mg/kg + Ipilimumab 3 mg/kg every three weeks (Q3W)(induction phase) followed by Nivolumab 480 mg every 4 weeks (Q4W)(consolidation phase) until unacceptable toxicity, disease progression (PD), investigator ́s decision, patient's consent withdrawal or death by any cause, whichever occurs first.

* Induction phase (Total of 4 cycles Q3W)

  * Nivolumab at 1 mg/kg by intravenous (IV) infusion on D1 of each cycle.
  * Ipilimumab at 3 mg/kg by intravenous (IV) infusion on D1 of each cycle.
* Consolidation phase (Cycles Q4W) ○ Nivolumab at a fixed dose of 480 mg by intravenous (IV) infusion on D1 of each cycle. The maximum duration of treatment with nivolumab will be 2 years, and patients will discontinue treatment at any time in case of unacceptable toxicity, disease progression (PD), investigator ́s decision, patient's consent withdrawal or death by any cause, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥ 18 years old.

2- Written informed consent approved by the Independent Ethics Committee (IEC), prior to the performance of any trial activities.

3- Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.

4- Histologically confirmed, unresectable locally advanced or metastatic transitional cell carcinoma of the urothelium.

* Also termed urothelial cell carcinoma [UCC] of the urinary tract; including renal pelvis, ureters, urinary bladder, and urethra).

  5- Stage IV disease (T4b, N0, M0; any T, N1-N3, M0; any T, any N, M1) at the start of first line chemotherapy.

  6- Prior first-line chemotherapy must have consisted of at least 4 cycles and no more than 6 cycles of gemcitabine plus cisplatin and/or gemcitabine plus carboplatin.

  7- Patient inclusion within the trial must occur within 3-12 weeks after the last dose of chemotherapy (3-12 weeks treatment-free interval).

  8- Only patients without progressive disease as per RECIST v1.1 guidelines after 4-6 cycles of chemotherapy will be allowed to be included. Baseline CT scan before inclusion should confirm that patients are on CR, PR or SD according to RECIST 1.1 criteria.

  9- Tumor tissue (formalin-fixed paraffin-embedded (FFPE) archival or recent acquisition) must be available at baseline.

Note: Fine Needle Aspiration [FNA] and bone metastases samples are not acceptable. If an insufficient amount of tumor tissue from an unresectable or metastatic site is available prior to the start of the screening phase, subjects must consent to allow the acquisition of additional tumor tissue. This may be discussed with the PI if a new biopsy is feasible.

10- Patients with adequate normal organ and marrow function as defined below:

1. Haemoglobin ≥ 9.0 g/dL.
2. Absolute neutrophil count (ANC) > 1500 per mm3.
3. Platelet count ≥ 100,000 per mm3.
4. Serum bilirubin ≤ 1.5 X institutional upper limit of normal (ULN) unless liver metastases are present, in which case it must be ≤ 2X ULN. This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of haemolysis or hepatic pathology); however, they will be allowed only in consultation with their physician.
5. Serum transaminases (ALT, AST and GGT) ≤ 2.5X institutional upper limit of normal unless liver metastases are present, in which case it must be ≤ 3X ULN.
6. Measured creatinine clearance (CL) > 30 mL/min or Calculated creatinine CL > 40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for the determination of creatinine clearance.

   11- Female subjects of childbearing potential (WOCBP) must provide a negative urine pregnancy test at screening, and must agree to use a medically accepted and highly effective birth control method (i.e. those with a failure rate less than 1%; refer to ANNEX III) for the duration of the study treatment and for 5 months after the last dose of study treatment.

A woman is considered of childbearing potential ( i.e. fertile) following menarche and until becoming post-menopausal unless permanently sterile. Women will be considered post-menopausal if they have been amenorrhoeic for 12 months without an alternative medical cause. The following age-specific requirements apply:

1. Amenorrheic for ≥1 year in the absence of chemotherapy and/or hormonal treatments
2. Luteinizing hormone (LH) and/or follicle stimulating hormone and/or estradiol levels in the post-menopausal range
3. Radiation induced oophorectomy with last menses >1 year ago
4. Chemotherapy induced menopause with >1 year interval since last menses
5. Surgical sterilization (bilateral oophorectomy or hysterectomy)
6. Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy)
7. Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

   12- Willingness and ability of patients to comply with the protocol for the duration of the study including undergoing treatment as well as availability for scheduled visits and examinations including follow up.

   Exclusion Criteria:
   1. ECOG performance status of >1 (Karnofsky < 70%).
   2. Patients whose disease progressed by RECIST v1.1 on or after first-line chemotherapy for urothelial cancer in the advanced or metastatic setting.
   3. Prior immunotherapy with IL-2, IFN-a or treatment with any immune checkpoint inhibitor therapy (e.g, CTLA4, PD-1, or PD-L1 targeting agent) for the unresectable metastatic setting.

      Note: Patients may have received immunotherapy in the adjuvant setting as long as the last dose of adjuvant was administered at least 12 months prior to the first dose of trial treatment.
   4. Receipt of any type of systemic chemotherapy or anticancer therapy within 3 weeks before starting treatment.
   5. Previously identified allergy or hypersensitivity to components of the study treatment formulations.
   6. History of allogeneic organ transplant.
   7. Any non-cancer treatment with vaccines used for the prevention of infectious diseases (up to 1 month before or after any dose of ipilimumab and nivolumab).
   8. Major surgery (i.e. cystectomy) less than 28 days prior to the first dose of study treatment.
   9. Patients with known symptomatic central nervous system (CNS) metastases requiring steroids. Patients with previously diagnosed CNS metastases are eligible if they have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to inclusion, have discontinued corticosteroid treatment for these metastases for at least 4 weeks, and are neurologically stable.
   10. Subjects that have a diagnosis of immunodeficiency or are receiving systemic steroid therapy or any other form of immunosuppressive therapy within 28 days prior to the first dose of trial treatment, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses (which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid).
   11. Active or prior documented autoimmune disease within the past 2 years which requires systemic therapy.

       Note: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded. Subjects with Type I diabetes mellitus are not excluded.
   12. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease and ulcerative colitis).
   13. Inadequate haematological/organ function.
   14. Any of the following in the previous 6 months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, deep vein thrombosis, or symptomatic pulmonary embolism.
   15. Persistence of any toxicities attributed to prior anti-cancer therapy, other than alopecia, that have not resolved to Grade 1 (NCI-CTCAE v5.0) or baseline before administration of study treatment.
   16. Active hepatitis B virus or hepatitis C virus.
   17. Vaccination within 4 weeks of the first dose of study treatment and while on trial is prohibited except for administration of inactivated vaccines (i.e. SARS-CoV-2 and Influenza vaccines will be permitted).
   18. Patients who have a known secondary malignancy that is progressing or has required active treatment within the past 2 years.

       Note: Patients with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ that have undergone potentially curative therapy are eligible.
   19. Pregnant or lactating females. Fertile and sexually active patients that are not willing to use the appropriate highly effective contraceptive methods.
   20. Any underlying medical or psychiatric disorder, which, in the opinion of the investigator, makes the administration of ipilimumab and nivolumab unsafe or interferes with the informed consent process or trial procedures.
   21. Participation in other studies involving investigational drug(s) within 4 weeks prior to inclusion. Observational studies are permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-07-06 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | Throughout the study period, approximately 12 months per patient from first study dose.
  PFS is defined as the time from the first dose of study treatment date until the first documentation disease progression or death from any cause, whichever occurs first. A subject who has not confirmed progression will be censored at the last known disease evaluation. Patients who have not progressed and start a new line of treatment will be censored at the date of the last adequate tumor assessment prior to starting the next line of therapy. Estimated by Kaplan Meier.
progression-free survival (PFS) in PL-D1 positive patients | Throughout the study period, approximately 12 months per patient from first study dose.
  subgroup analysis of PFS. Same definition of PFS as Outcome 1 applies.

SECONDARY OUTCOMES:
Overall Survival (OS) | Throughout the study period, approximately 12 months per patient from first study dose.
  Time from the first dose of study treatment date to the date of death and the proportion/percentage of patients alive at the end of follow-up. A subject who has not died will be censored at the last known date alive. Estimated by Kaplan Meier
Clinical benefit rate (CBR) | Throughout the study period, approximately 12 months per patient from first study dose.
  Percentage/proportion of patients with complete response (CR) or partial response (PR), according to ORR definition for the trial, or maintained stable disease (SD) as their overall best response throughout the study period, assessed by imaging follow-up (CT scan/MRI) and RECIST 1.1 criteria. Stable disease should be maintained for at least 4 months to be considered as a CBR event.
Duration of response (DoR) | Throughout the study period, approximately 12 months per patient from first study dose.
  Time from first confirmed response (CR or PR), according to ORR definition for the trial, to the date of the documented PD as determined using RECIST 1.1 criteria or death due to any cause, whichever occurs first.
Post-chemotherapy PFS (cPFS) | Throughout the study period, approximately 12 months per patient from first study dose.
  defined as the time from first dosing date of chemotherapy until the first documentation disease progression or death from any cause, whichever occurs first.
Post-chemotherapy OS (cOS) | Throughout the study period, approximately 12 months per patient from first study dose.
  Time from first dosing of chemotherapy date to the date of death and the proportion/percentage of patients alive at the end of follow-up.
Frequency of adverse events | Throughout the study period, approximately 12 months per patient from first study dose.
  Number of patients experiencing adverse events from the total of patients exposed to study drug
Frequency of treatment-related adverse events | Throughout the study period, approximately 12 months per patient from first study dose.
  Number of patients experiencing adverse events related to the study treatment from the total of patients exposed to study drug
Quality of life (QoL) patient reported outcomes | Throughout the study period, approximately 12 months per patient from first study dose.
  Patient reported outcomes assessed through the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ-C30), version 3 and the EuroQoL five-dimensions, 5 level (EQ- 5D-5L) questionnaire. Median scores for both questionnaires will be provided.
Objective response rate (ORR) | Throughout the study period, approximately 12 months per patient from first study dose.
  Assessed by the investigator by imaging follow-up (CT scan/MRI) using the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. This will be considered as the percentage/proportion of patients with confirmed complete response (CR) or partial response (PR) as their overall best response throughout the study period. Objective responses will be assessed by the investigator according to the Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo de Velasco, Study Chair — Hospital Universitario 12 de Octubre
Locations (12):
- Spain (12):
  - Hospital Universitario Juan Ramón Jiménez, Huelva, Andalusia
  - Hospital Universitario Virgen de la Macarena, Seville, Andalusia
  - Hospital Clínico Universitario de Zaragoza, Zaragoza, Aragon
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Complejo asistencial universitario de Salamanca, Salamanca, Castille and León
  - Hospital Universitario de Toledo, Toledo, Castille-La Mancha
  - Hospital Clínic de Barcelona, Barcelona, Catalonia
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela, Galicia
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario de la Ribera, Alzira, Valencia

IPD SHARING:
Plan to Share IPD: No